CLINICAL TRIAL: NCT01627457
Title: Heart Cycle Prestudy Guided Exercise (GEx) for Coronary Artery Disease Patients (CAD) "GEx Home Application Testing"
Brief Title: Heart Cycle Prestudy
Acronym: PreGEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-094
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction
Keywords: Coronary Artery Disease; Guided Exercise System including ECG Vest with vital signs sensors and PDA; Validation Telemedical Device in regard to accuracy and safety of data; Homely Rehabilitation; Practicability and technical problems at home
MeSH Terms: conditions — Coronary Artery Disease; Ductus Arteriosus, Patent | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GEx Training (Experimental): CAD Patients in cardiac rehabilitation phase II (inpatient) and phase III (at home)in order to analyze data for quality of heart rate measurement and data acquisition by device as well as for practicability and technical problems at home.
  Interventions: Device: Guided Exercise (GEx) system

INTERVENTIONS:
Device: Guided Exercise (GEx) system — 30 CAD patients will wear the GEx system while they are trained during inpatient cardiac rehabilitation (phase II) in order to evaluate accuracy and safety of data like heart rate, breathing, ECG three times a week for about three weeks. In a second step these patients train at home (phase III) in order to evaluate practicability and technical problems of the GEx device three times a week for about three weeks.

SUMMARY:
In this Prestudy which will be followed by the multicentral GEx- main-trial, the feasibility of a new cardiac rehabilitation device (GEx system) is proved with coronary heart disease patients who participate in cardiac rehabilitation training exercise at the rehabilitation clinic (phase II) and subsequently at home (phase III). The GEx system consists of a easy-to-wear vest with integrated electrodes to measure electrocardiogram (ECG), respiration and activity, furthermore of a PDA to collect and store the monitored data and a cradle to charge the batteries. Several physiological parameters are extracted from thes measured vital signs like heart rate, breathing rate, ECG and activity. In this pretrial first the GEx sensor system is validated during guided exercise of the patients in the rehabilitation clinic (phase II). Subsequently at home (phase III) the practicability of the vest and sensors and possible technical problems in real- life use are proved. This means after moderate training like walking, cycling or running at home for 3 weeks patients will report the feasibility of usage. The ECG data and breathing- frequency data will be analyzed to see if data are recorded and transmitted well in regard to technical problems.

DETAILED DESCRIPTION:
During the rehabilitation process (phase II) of patients with coronary heart disease (CAD) 30 patients are recruited and are made familiar with the new Guided Exercise (GEx) training system during exercise training; they are supervised and provided with training instructions by a medicine for 3 times a week 3 weeks long. At the beginning and at the end of the study the patient has to undergo several tests of the clinical routine such as a cardiopulmonary test (CPX), echocardiography and lactate measurement;additionally, this test will be registered by the system to obtain information about the detection of heart rate rise for example. Data will be analyzed for quality of heart rate measurement and data acquisition by the device.

In a second step the GEx system is handed to these 30 patients when they leave in-patient cardiac rehabilitation (CR). The pre-trial serves to gather information about the practicability and technical problem during real-life use. Therefore at home these 30 patients will continue with moderate endurance training like walking, cycling or running while wearing the GEx system three times a week for 3 weeks. After three weeks patients will come back to the clinic to undergo the end examination and to report the feasibility of usage. The ECG data and breathing frequency data will be analyzed to see if data are recorded and transmitted well in regard to technical problems.

If accurate and safe data are received the following GEx- main- trial (ID 11-020) will investigate the GEx- system for CAD patients in regard to improvement of physical capacities obtained in long term adherence to home based rehabilitation programs (phase III) including feedback to patients compared to national standard rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from CAD and presenting after an acute myocardial infarction or elective coronary intervention
* Patients willing to exercise
* With a preference for walking/ cycling/ running
* Eligible for the normal local rehabilitation program
* Contractually capable and mentally able to understand and follow the instructions of the study personnel
* Able to give informed consent

Exclusion Criteria:

* Ejection Fraction at discharge from hospital < 30%
* Unwillingness or lack of capability to handle the device
* Unable to perform exercise
* Severe congestive heart failure NYHA III/IV
* Severe valve disease without replacement
* Slow healing wounds
* Women who are pregnant or breastfeeding
* Refusal of device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of accuracy and safety of data of the GEx system received during in-patient cardiac rehabilitation (phase II) and evaluation of practicability and technical problems in real- life use during cardiac rehabilitation at home (phase III). | 6 Months
  The GEx system is evaluated during in-patient cardiac rehabilitation supervised by cardiologists in order to analyze data for quality of heart rate measurement and data acquisition by device. 30 Patients undergo moderate training exercise like walking, cycling or running three times a week three weeks long. In a second step practicability and technical problems are tested during continuation of the moderate training of the patient at home. The Evaluation is performed by CPX, lactate measurement, 2D-Echo, questionnaires and device data like heart rate and breathing rate.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schauerte, Professor MD, Principal Investigator — University Hospital Aachen, Department of Cardiology
Locations (1):
- Medical Clinic I, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany